CLINICAL TRIAL: NCT03930420
Title: Training Local Health Departments to Disseminate Evidence-Based Interventions to Small and Low-Wage Worksites
Brief Title: Training LHDs to Disseminate Evidence-Based Interventions to Small Worksites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Association of Chronic Disease Directors (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peggy Hannon, Professor: School of Public Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004627; 2R01CA160217 (NIH); NCI-2021-02876 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1121453 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Health Behavior
Keywords: evidence-based practice; implementation science; public health practice
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: The research team will use a hybrid type III study design to conduct a randomized controlled trial (RCT) comparing the effect of standard Connect to Wellness training and TA to the effect of training plus enhanced TA on primary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): Local health department staff in the standard arm will receive Connect to Wellness intervention materials, multiple real-time training sessions delivered via webinar, access to a web-based platform that includes all intervention and training materials and has features allowing them to communicate with each other and with research staff, and a monthly group technical assistance call.
  Interventions: Behavioral: Connect to Wellness
- Enhanced (Experimental): Local health department staff in the enhanced arm will receive all the Connect to Wellness intervention materials, training, and support as described for the standard arm. In addition, the participants in the enhanced arm can telephone research staff at will to receive additional technical assistance. Research staff will also contact participants monthly, if they do not request assistance proactively.
  Interventions: Behavioral: Connect to Wellness

INTERVENTIONS:
Behavioral: Connect to Wellness — The research team will train LHD staff and offer them technical assistance to work with small worksites. LHD staff will be trained to deliver the Connect to Wellness program to worksites. Connect to Wellness is a program to disseminate EBIs to small worksites. Worksites receive guidance about EBIs and ongoing implementation assistance from a trained interventionist. In this study, LHD staff will be the interventionists. Worksites participating in Connect to Wellness complete three phases of activities, Assessment, Recommendations, and Implementation. LHD staff will receive Connect to Wellness intervention materials, multiple webinars delivered in real-time, access to a comprehensive intervention and training platform with features that allow them to connect with each other and with research staff, and group technical assistance calls to support their ability to recruit worksites in their communities and deliver Connect to Wellness to these worksites.

SUMMARY:
The proposed project will advance implementation science by comparing the effectiveness of different levels of technical support in an important but understudied community-based setting: local health departments. The proposed project will also bring Connect to Wellness, an evidence-based approach to disseminating evidence-based interventions and providing implementation support to small worksites, to 40 local health departments and worksites in their communities across the United States. Findings will identify the best approach for national scale-up of Connect to Wellness.

DETAILED DESCRIPTION:
Cancer and other chronic diseases are the leading causes of death in the United States for working-age adults. There are several behavioral risk factors that increase disease risk, including missed cancer screenings, physical inactivity, poor eating habits, and tobacco use. Evidence-based interventions (EBIs) exist that improve each of these risk behaviors, and many of these EBIs can be implemented in worksites where the majority of U.S. adults spend most of their waking hours. There are significant disparities in access to worksite EBIs; large worksites (more than 1000 employees) are much more likely to offer EBIs to their employees than small worksites with less than 250 employees. The American Cancer Society (ACS) and the University of Washington Health Promotion Research Center (HPRC) developed Connect to Wellness, a package of EBIs appropriate and feasible for small worksites. A recent randomized controlled trial of Connect to Wellness with 69 small worksites showed that worksites in the Connect to Wellness arms implemented significantly more EBIs at follow-up than worksites in the delayed control arm.

The objective of the present study is to test different methods of scaling up Connect to Wellness. Local health departments (LHDs) cover almost every community in the United States and most LHDs' missions include preventing chronic disease. In a separate project, UW pilot-tested training staff in six LHDs in Washington State to deliver Connect to Wellness to worksites in their communities. LHD staff completed the training and recruited worksites to participate in Connect to Wellness; these worksites implemented EBIs. The primary goals of this competing renewal are (a) to scale up Connect to Wellness by training staff in LHDs across the United States to deliver Connect to Wellness to small employers in their communities, and (b) to further implementation science by conducting a hybrid type III trial comparing the effectiveness and costs of two different implementation strategies. These goals will be achieved through three specific aims, guided by the HPRC Dissemination and Implementation Framework. The research team will conduct qualitative audience research with state and local health department directors and local health department staff to refine training and support approaches (Aim 1); conduct a hybrid type III trial comparing standard and enhanced technical assistance combined with online training for Connect to Wellness (Aim 2); and measure the costs of each strategy, both to the local health departments and to the research team (Aim 3). The proposed activities will increase the reach of Connect to Wellness across the United States to small employers with limited capacity for and access to EBIs. These activities will also advance implementation science by measuring the impact and costs of implementation strategies offering different levels of ongoing support. The findings from this project may inform implementation strategies for other workplace health promotion programs focused on EBIs and small worksites, as well as a variety of implementation efforts that include partnerships with LHDs. Aim 2 and Aim 3 activities will be achieved through the randomized trial described in the protocol registered on ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Staff in local health departments in United States (50 states and District of Columbia)
* Local health department willing to support one or more staff to participate for 24 months
* Local health department willing to attempt to recruit 15 or more worksites to participate in Connect to Wellness over 24 months
* Able to speak and read English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Hannon, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team is committed to making the data collected available to other scientists and the public after a reasonable period of time for main analyses and the publication of results. The data and the related documentation will be archived at the Health Promotion Research Center and will be available (in a de-identified format) upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available starting in May 2024.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Health departments
Period: Overall Study
Arm/Group | Standard | Enhanced
Started | 31; 10 Health departments | 38; 11 Health departments
Completed | 24; 8 Health departments | 29; 7 Health departments
Not Completed | 7; 2 Health departments | 9; 4 Health departments
Not completed — Withdrawal by Subject | 7 | 9

BASELINE CHARACTERISTICS:
Population: These numbers are smaller than the participant flow numbers because some staff did not provide data about their age, race, or gender
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard | Enhanced | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 25 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 13 | 21 | 34
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Worksites
Description: The outcome measure is the average number of worksites recruited by the health departments
Time Frame: 24 months
Population: We randomized at the level of health departments, as we recruited health departments to participate in the study and trained their staff to deliver Connect to Wellness. Thus, health departments are the unit of analysis.
Measure: Mean (Full Range); unit: Worksites
Units Other Than Participants: Local health departments
Arm/Group | Standard | Enhanced
Number analyzed (Participants) | 31 | 38
Number analyzed (Local health departments) | 10 | 11
Worksites
  Number of worksites at baseline | 0 [0 to 0] | 0 [0 to 0]
  Number of worksites at 24 months | 1.2 [0 to 6] | 1 [0 to 4]

2. Primary Outcome: Worksite EBI Implementation
Description: The evidence-based intervention implementation score for each worksite that participates in the Connect to Wellness intervention; possible score range is 0-100, with higher numbers reflecting higher EBI implementation.
Time Frame: Baseline
Population: Health departments were generally unable to collect follow-up outcome data from the worksites they delivered Connect to Wellness to; only 3 worksites provided follow-up data and these were all in a single study arm. For this reason, even though we planned to collect follow-up data at 12 months, we present only worksites' baseline EBI implementation scores.
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: Local health departments
Arm/Group | Standard | Enhanced
Number analyzed (Participants) | 31 | 38
Number analyzed (Local health departments) | 10 | 11
score on a scale | 35 [17 to 59] | 22 [7 to 70]

ADVERSE EVENTS:
Description: Death, serious adverse events, and other non-serious adverse events were not assessed for the study.
Arm/Group | Standard | Enhanced
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study started at the onset of the COVID-19 pandemic; this was an overwhelming barrier to completing study activities for our health department partners. Those that participated were committed to the research goals, but most were unable to meet recruitment or data collection needs. We did additional research with health departments to better understand these barriers, and with employers/employees to identify post-pandemic workplace health needs of small, low-wage businesses and employees.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03930420/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT03930420/SAP_001.pdf